CLINICAL TRIAL: NCT03830229
Title: Long Term Follow-up of Mesothelioma Patients and Their Family Members With Germline Mutations in BAP1 and Other Genes
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190049; 19-C-0049
Record Dates: First submitted 2019-02-02; First posted 2019-02-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12-17

CONDITIONS: Mesothelioma; Families
Keywords: DNA Repair Genes; Natural History
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Germline positive mesothelioma: Individuals with mesothelioma who have a BAP1 or other DNA repair/cancer predisposition mutation regardless of CLIA (or equivalent) confirmation
- 2/CLIA confirmed germline mutation without mesothelioma: Individuals with a CLIA (or equivalent) confirmed BAP1 or other DNA repair/cancer predisposition mutation who do not have a diagnosis of mesothelioma

SUMMARY:
Background:

-A gene provides instructions to the body. Mutated genes can sometimes cause cancer. Germline mutations are those people are born with. These mutations in the BAP1 gene can cause mesothelioma and other cancers. Researchers want to study people with germline mutations of BAP1 and other genes known to cause cancer.

Objective:

-To learn how cancer might develop in people with certain gene mutations.

Eligibility:

-People ages 2 and older with a germline mutation in BAP1 or another gene that might cause cancer

Design:

* Participants will be screened with:

  * Medical and family history
  * Saliva test
* Participants with mesothelioma will be in the NIH Group. Participants without mesothelioma can choose to be in either the NIH Group or the Remote Group.
* Remote Group participants will have a medical and family history by phone. If they have tumor tissue from a previous surgery, it will be tested. They will be contacted once a year by phone.
* NIH Group participants will have a baseline visit. This can take up to 4 days. They may have to stay in the area overnight. The visit will include:

  * Physical exam
  * Evaluation of tumor tissue if available
  * Optional tumor biopsy
  * Blood tests
  * Scans: A machine will take pictures of the body.
  * Photographs of skin lesions or other issues
  * Skin exam
  * Eye exam
* NIH Group participants will have visits once or twice a year. These will include a physical exam, lab tests, scans, and other tests as needed.
* Participants who have a confirmed mutation will be asked to contact any relatives who may be at risk and ask them about joining the study.

DETAILED DESCRIPTION:
Background:

* BRCA1-Associated Protein-1 (BAP1), a deubiquitinase involved in regulating DNA repair enzymes, is believed to be a prominent mutation in malignant mesothelioma
* Germline mutations involving BAP1 have been reported in familial studies. These have been associated with a higher likelihood of mesothelioma as well as several other malignancies, including uveal melanoma, cutaneous melanomas, renal cell carcinoma and cholangiocarcinoma
* BAP1 mutations, if found, have a high probability of detecting multiple malignancies in family members.

Objectives:

-To characterize the natural and clinical history of malignant mesothelioma patients and their family members who have germline mutations in BAP1 and other DNA repair/cancer predisposition genes

Eligibility for Genetic Testing:

Cohort 1

-Individual with mesothelioma with deleterious germline mutations in BAP1 or another DNA-repair/cancer predisposition gene(s) (previous testing may have been research or clinical)

OR

* Individual with a diagnosis of mesothelioma who is otherwise eligible for testing on Cohort 2
* Age greater than or equal to 2

Cohort 2

-Individual with a germline BAP1 mutation who does not have a history of mesothelioma (previous testing may have been research or clinical)

OR

-Individual with no personal history of mesothelioma with:

--a first degree biological relative (living or deceased) with a history of mesothelioma

OR

--a first degree biological relative with a CLIA (or equivalent) confirmed germline mutation in BAP1

OR

--a second degree biological relative with a CLIA (or equivalent) confirmed germline mutation in BAP1 if relevant first degree relative is deceased or unavailable for testing

OR

--a first degree biological relative with mesothelioma and a CLIA (or equivalent) confirmed germline mutation in another DNA-repair/cancer predisposition genes

OR

--a second degree biological relative with mesothelioma and a CLIA (or equivalent) confirmed germline mutation in BAP1

-Age greater than or equal to 16 unless participant has a BAP1 mutation or a first degree biological relative with a confirmed TP53 or BAP1 germline mutation; in such cases, will begin screening at age greater than or equal to 2

Eligibility for Surveillance:

Cohort 1

-No additional criteria

Cohort 2

-Testing performed on study must confirm presence of germline mutation in BAP1 or another DNA repair/cancer predisposition gene(s)

Design:

* Individuals with suspected hereditary predisposition to mesothelioma and their families will be recruited to assess for genetic mutations, and to study the natural history of malignancies occurring in germline BAP1 mutations as well as other mutations involved in DNA repair.
* Screening examinations will be offered to those with germline BAP1 mutations as well as other mutations involved in DNA repair/cancer predisposition.
* We will determine if there is a relationship between germline mutation and disease phenotype.

ELIGIBILITY:
* Inclusion Criteria:

Inclusion Criteria for Genetic Testing:

Cohort 1:

* Participant with pathology confirming a diagnosis of mesothelioma.
* Participant must have a deleterious germline BAP1 mutation. Results from either research or clinical analyses are sufficient for this criterion.

OR

-Participant with mesothelioma otherwise eligible for genetic testing in Cohort 2

OR

* Participant must have deleterious germline mutation in another DNA repair/cancer predisposition gene(s) that is listed on a commercially available, cancer-associated common or customized gene panel. Results from either research or clinical analyses are sufficient for this criterion.
* Age greater than or equal to 2 years

Cohort 2:

-Individual with a germline BAP1 mutation who does not have a history of mesothelioma (other cancers are allowed). Results from either research or clinical analyses are sufficient for this criterion.

OR

-Individual with no history of mesothelioma with:

--A biological first degree relative (living or deceased) with a history of mesothelioma

OR

--A first degree biological relative with a CLIA (or equivalent) confirmed germline mutation in BAP1

OR

--A second degree biological relative with a CLIA (or equivalent) confirmed germline mutation in BAP1 if relevant first degree relative is deceased or unavailable for testing,

OR

--A first degree biological relative with mesothelioma and a CLIA (or equivalent) confirmed germline mutation in another DNA-repair/cancer predisposition gene that is listed on a commercially available, cancer-associated common or customized gene panel

OR

* A second degree biological relative with mesothelioma and a CLIA (or equivalent) confirmed germline mutation in BAP1

  -Age:
* greater than or equal to 2 years for participants with a BAP1 or TP53 mutation or with a first degree relative that has a germline mutation in TP53 or BAP1
* greater than or equal to 16 years for all other eligible potential mutations

All participants must understand and be willing to sign a written informed consent

Exclusion Criteria for Genetic Testing

None

Inclusion Criteria for Surveillance:

* Genetic testing criteria including age restrictions for respective cohorts must be met
* Participants in Cohort 1 may be enrolled with positive results for germline BAP1 mutation or another DNA repair/cancer predisposition gene(s) that is listed on a commercially available, cancer-associated common or customized gene panel regardless of CLIA (or equivalent) confirmation
* Participants in Cohort 2 must have CLIA (or equivalent) confirmed germline BAP1 mutation or another DNA repair/cancer predisposition gene(s) that is listed on a commercially available, cancer-associated common or customized gene panel

OR

-if germline status negative, have a biological relative that is enrolled for surveillance

Exclusion Criteria for Surveillance:

None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with mesothelioma and family members as well as individuals with CLIA documented germline BAP-1 and other DNA repair/cancer predisposition mutations
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2027-07-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and frequencies of Cancers | ongoing
  Standard exploratory and descriptive measures will be used. Counts, incidence, and frequencies of cancers identified via screening procedures on this trial will be reported, all in the context of an exploratory study with appropriate caveats.

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data in BTRIS will be shared throughout the course of the study and indefinitely with the permission of the investigator.@@@@@@Genomic data will be shared from the time of upload to dbGaP.
Access Criteria: Clinical IPD will be shared through the BTRIS database for open ended analysis. All BTRIS subscribers, generally limited to the NIH Clinical Center, may request data.@@@@@@Genomic IPD will be shared through dbGaP, per rules of the database, for purposes of genomic analysis.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0049.html